CLINICAL TRIAL: NCT00840996
Title: Effect of Perioperative Intravenous Lidocaine Administration or Epidural Anesthesia on Postoperative Outcomes in Complex Spine Surgery
Brief Title: Perioperative Intravenous Lidocaine or Epidural Anesthesia on Outcomes in Complex Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ehab Farag, Ehag Farag, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-209; NCT00706524 (obsolete NCT alias)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-10

CONDITIONS: Spine Surgery
Keywords: Spine Surgery; Intraocular pressure; Lidocaine; Epidural Anesthetic
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Perioperative placebo IV infusion besides the standard anesthesia care, including general anesthesia and postoperative patient controlled analgesia.
  Interventions: Drug: placebo
- Lidocaine (Active Comparator): Perioperative intravenous lidocaine infusion besides the standard anesthesia care, including general anesthesia plus and post operative patient controlled analgesia.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — perioperative intravenous lidocaine (2 mg/kg/h) with maximum of 200 mg/h starting at induction of anesthesia and continuing until discharge from the PACU or a maximum of 8 hours
  Other Names: Liodocaine
  Arms: Lidocaine
Drug: placebo — perioperative placebo IV saline infusion of 2 mg/kg/h with maximum of 200 mg/h starting at induction of anesthesia and continuing until discharge from the PACU or a maximum of 8 hours
  Arms: Placebo

SUMMARY:
The purpose of this study is determine if epidural anesthesia administered after surgery or lidocaine administered during surgery will decrease inflammation after spinal surgery and decrease the need for post operative pain medication compared to intravenous patient controlled analgesia. Participants undergoing spine surgery will be randomized into one of two groups;

- A.) General Anesthesia and postoperative Patient Controlled Analgesia and placebo IV infusion.

B.) General Anesthesia plus perioperative intravenous lidocaine infusion, and post operative Patient Controlled Analgesia.

DETAILED DESCRIPTION:
According to a survey of 1570 U.S neurosurgeons, in the United States about 527.000 spine surgeries were done in 1999. This represents close to 65% of the procedures performed by neurosurgeons. Furthermore, the number of hospitalizations related with spine surgery has significantly increased since 1970.

IV PCA is considered the standard of care for postoperative pain control after surgery. Intravenous opioids have significant side effects such as respiratory depression, postoperative nausea and vomiting and sedation. Furthermore, they cause delayed return of bowel function and ileus.

There is the possibility of surgically inserting a catheter into the epidural space at the end of surgery. In general epidural analgesia provides excellent pain relief after surgery and decreases opioid consumption significantly und thus opioid related postoperative complications. Furthermore epidural anesthesia affects the surgical stress response and might decrease inflammatory responses after surgery, thereby improving postoperative recovery and mobilization of the patients.

Intravenous local anesthetics have potent anti-inflammatory properties. They also decrease postoperative opioid consumption. Clinical studies have shown that perioperative local anesthetic administration significantly reduces the incidence of thrombosis and postoperative pain, shortens postoperative ileus and decreases duration of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years old at time of surgery - adult patients differ from pediatric patients in that adult spines are stiffer than pediatric patient.
* Elective spine surgery
* Two levels laminectomies or above with or without fusion or instrumentatioN
* General anesthesia
* Surgery performed at Cleveland Clinic with informed consent signed prior to sedation or anesthesia - consistent surgical team

Exclusion Criteria:

* contraindication to lidocaine such as substantial hepatic impairment (ALT or AST more than twice normal)
* renal impairment (serum creatinine >2 mg/dl),
* seizure disorder requiring medication within 2 years
* planned epidural anesthesia or analgesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Farag, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: With approval of the institutional review board at the Cleveland Clinic and written informed consent, between September 2009 to October 2011 we enrolled 116 patients to undergo elective multi-level spine surgery At Cleveland Clinic, Cleveland, Ohio, USA .
Groups:
- Placebo: Perioperative equal volume of saline placebo IV infusion
Period: Overall Study
Arm/Group | Lidocaine | Placebo
Started | 58 | 58
Completed | 57 | 58
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine | Placebo | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11) | 54 (11) | 56 (11)
Gender [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Scores
Description: The pain score as measured by verbal response scores (scale ranging from 0 to 10 with 0=no pain; 10=worst pain) every 30 minutes during post anesthesia care unit stay, then per nursing floor protocol (roughly every 4-6 hours).
Time Frame: From admission to the post anesthesia care unit through postoperative day 2 (or discharge, if earlier).
Measure: Mean (Standard Deviation); unit: verbal response scores
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 57 | 58
verbal response scores | 4.4 (0.13) | 5.3 (0.13)
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; Postoperative analgesia was characterized using both pain scores and opioid consumption .We considered one of the groups to be better than the other on postoperative pain control with superiority on either outcome, in the presence of noninferiority on both outcomes. Thus, our primary hypothesis was assessed in a joint hypothesis testing framework; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Test for superiority adjusted for 2 primary comparisons (2 outcomes); Llinear mixed-effects accounts for correlation exhibited by the repeated pain measurements on a given patient (spatial power correlation structure); Mean Difference (Final Values) = -0.80, 97.5% CI 2-sided [-1.23 to -0.40]

2. Primary Outcome: Opioid Medication Requirement, mg in IV Morphine Equivalent
Description: Opioid consumption during the initial 48 postoperative hours was converted to IV morphine sulfate equivalents
Time Frame: through postoperative day 2 (or discharge, if earlier)
Measure: Mean (Standard Deviation); unit: mg IV morphine equivalent
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 57 | 58
mg IV morphine equivalent | 55 (8) | 74 (11)
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority margin: ratio of the geometric means not more than 1.3 greater (mean mg IV morphine equivalent not more than 30% greater ) than that of the other group; p = 0.011, Regression, Linear — Noninferiority hypotheses were evaluated against a one-sided significance criterion of 0.025 [adjusting for testing in both directions: lidocaine vs. control and vs. control vs. lidocaine ]; Log-linear regression model was used; 0.1 mg added before taking the logarithm to accommodate the 2 patients who received 0 mg opioids; the ratio of the geometric means = 0.8, 95% CI 2-sided [0.65 to 1.21]

3. Secondary Outcome: Number of Participants With Any Major 30-day Post Operative Complications
Description: The occurrence in an individual of one or more the following major complications, including pneumonia, respiratory failure, prolonged use or need for reinsertion of chest tube, cardiac arrest, arrhythmia, congestive heart failure, stroke, intravascular coagulopathy, thromboembolic disease (pulmonary embolism), injury to great vessels, delirium, monoplegia or paraplegia, upper gastrointestinal bleeding, gastrointestinal block, ureteral obstruction, syndrome of inappropriate antidiruretic hormone secretion, wound infection requiring debridement, sepsis, and readmission.
Time Frame: 30 days after surgery
Measure: Number; unit: participants
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 57 | 58
participants | 2 | 5
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; Test type: Superiority or Other; p = 0.049, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.84 to 1.00]

4. Secondary Outcome: Postoperative Nausea and Vomiting (PONV)
Description: Postoperative Nausea and Vomiting (PONV)will be noted during day one and day two postoperative.
Time Frame: post op day one and two or till hospital discharge
Population: We only have 39 and 36 patients for comparison of PONV at day two after surgery, since the rest were discharged by that time
Measure: Number; unit: participants
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 39 | 36
participants
  Nausea | 4 | 8
  Vomiting | 2 | 1
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; Nausea - POD 2; Test type: Superiority or Other; p = 0.31, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.77 to 1.09]
Statistical Analysis 2: Comparison: Lidocaine vs Placebo; Vomiting - POD 2; Test type: Superiority or Other; p = 0.44, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.94 to 1.14]

5. Secondary Outcome: Duration of Hospitalization
Description: Length of hospital stay will be recorded in days.
Time Frame: At discharge
Population: 3 patients in the placebo group did not have duration of hospital stay recorded.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 57 | 55
days | 3 [2 to 4] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; Test type: Superiority or Other; p = 0.15, Regression, Linear; Mean Difference (Final Values) = -1, 95% CI 2-sided [-2.4 to 0.4]

6. Secondary Outcome: 12-item Short Form Survey (SF-12) Physical Health Composite Score
Description: Physical health composite score ranges from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: 30 days post operative
Population: Include the participants who finished the Acute SF 12 health survey at 30 days follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 54 | 55
units on a scale | 38 [31 to 47] | 33 [27 to 42]
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; Test type: Superiority or Other; p = 0.002, Regression, Linear; Mean Difference (Final Values) = 6.2, 95% CI 2-sided [2.3 to 10]

7. Secondary Outcome: 12-item Short Form Survey (SF-12) Physical Health Composite Score
Description: as for outcome 6
Time Frame: 90 days post operative
Population: Include the participants who finished the Acute SF 12 health survey at 90 days follow-up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lidocaine | Placebo
Number analyzed (Participants) | 51 | 54
units on a scale | 39 [31 to 49] | 34 [28 to 44]
Statistical Analysis 1: Comparison: Lidocaine vs Placebo; Test type: Superiority or Other; p = 0.04, Regression, Logistic; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [0.3 to 8.9]

ADVERSE EVENTS:
Arm/Group | Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/58
Other Adverse Events (participants affected / at risk) | 0/57 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No